CLINICAL TRIAL: NCT01485081
Title: Assessment of the Safety and Efficacy of the Danubio Paclitaxel-Eluting Balloon for the Treatment of Side Branches of de Novo Bifurcation Lesions in Native Coronary Arteries.
Brief Title: Safety and Efficacy Study of the DANUBIO Paclitaxel Eluting Balloon in Side Branches of de Novo Bifurcation Lesions (DEBSIDE)
Acronym: DEBSIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MINVASYS (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIN1101
Record Dates: First submitted 2011-11-14; First posted 2011-12-05 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Disease
Keywords: Bifurcation; Drug-eluting balloon; Paclitaxel-eluting balloon; Angioplasty; Coronary artery disease; Coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Danubio (Experimental)
  Interventions: Device: Danubio paclitaxel-eluting balloon

INTERVENTIONS:
Device: Danubio paclitaxel-eluting balloon — Inflation of the Danubio Paclitaxel Eluting Balloon in the side branch of a de novo bifurcation lesion.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the Danubio Paclitaxel Eluting Balloon for the treatment of side branches of de novo bifurcation lesions in native coronary arteries.

DETAILED DESCRIPTION:
The DEBSIDE clinical trial is a prospective, non-randomized, multicenter, interventional study evaluating the investigational Danubio Paclitaxel Eluting Coronary Balloon for the treatment of Side Branches (SB) of de novo bifurcation lesions with a side branch reference vessel diameter ≥2.0 mm and ≤3.0 mm. During the procedure, a dedicated drug-eluting bifurcated stent will be implanted in the main branch. The trial will allow the treatment of lesion of all Medina type except (0,0,1) in native coronary arteries with sequential predilatation of the main and side branch.

The DEBSIDE clinical trial will enroll 60 patients. All patients will receive Quantitative Coronary Angiography (QCA) before and after Drug-Eluting Balloon (DEB) inflation and at 6 months follow-up. All patients will have a clinical follow-up at 1, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. De novo bifurcation lesions following the Medina classification except (0,0,1).
2. Reference diameter main branch >= 2.5 and ≤ 3.5 mm and side branch >= 2.0 and ≤ 3.0 mm.
3. Main branch lesion length ≤ 26mm and side branch lesion ≤ 6mm.

   * For a 24mm stent in the main branch: main branch lesion length ≤ 14mm proximal and ≤ 12mm distal to the carina.
   * For a 18mm stent in the main branch: main branch lesion length ≤ 8mm proximal and ≤ 12mm distal to the carina.

   Indeed an additional stent (Amazonia PAX 8mm) can be overlapped distally with the Nile PAX if a target lesion segment ≤4mm remains uncovered after implantation of the bifurcated stent.
4. Maximum two bifurcation lesions per patient on two different vessels with at least one lesion treated with the procedure described on the protocol (involving the Danubio).
5. The side branch of the bifurcation involving the target lesion must be treated with the trial device (Danubio).
6. During the index procedure, in case of:

   * Treatment of a lesion in a vessel other than the target vessel or,
   * Treatment of a lesion in the target vessel distal to the target bifurcation lesion, The treatment of the non-target lesion must be successfully performed with a Drug-Eluting Stent before the treatment of the target lesion (residual stenosis <30%; stent well deployed; no residual dissection; normal TIMI flow; no chest pain; ECG unchanged compared to pre-procedural ECG).
7. Successful sequential main branch and side branch predilatation with a conventional balloon providing good angiographic result (i.e. absence of dissection, TIMI > III).
8. The patient is at least 18 years of age.
9. Non menopausal women must provide a negative pregnancy test and use a double contraception until the end of the study.
10. The patient has clinical evidence of ischemic heart disease, stable or unstable angina with signs of ischemia, silent ischemia, or a positive functional test.
11. The patient is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergent coronary artery bypass graft (CABG) surgery.
12. The patient or patient's legal representative has been informed of the nature of the trial and agrees to its provisions and has provided written informed consent as approved by the Ethics Committee (EC).
13. The patient agrees to return to the same research facility for required angiographic post-procedure follow-up visit at 6 months

Exclusion Criteria:

1. De novo bifurcation lesion Medina (0,0,1).
2. Left main bifurcation.
3. The Danubio covers beyond the side branch lesion distally with <2mm.
4. The stent covers beyond the main branch lesion proximally and distally with <2mm.
5. Heavily calcified lesions.
6. Severe tortuous lesions.
7. Evidence of extensive thrombosis or dissection within target vessel before the intervention
8. Documented left ventricular ejection fraction (LVEF) <30% at most recent evaluation.
9. Main branch of the target lesion stented with other device than Nile PAX.
10. Dissection or required additional treatment in the main or side branch of the target lesion after main branch stent implantation.
11. Untreated significant lesion >50% diameter stenosis remaining proximal or distal to the target lesion
12. A known hypersensitivity or contraindication to aspirin, heparin or bivaluridin, ticlopidine or clopidogrel, paclitaxel or drugs in similar class, cobalt chromium alloys, contrast media, which cannot be adequately pre-medicated.
13. Chronic total occlusion (CTO).
14. A serum creatinine level >2.0mg/dL within seven days prior to index procedure.
15. Evidence of an acute MI within 72 hours of the intended index procedure (according to ARC definition).
16. Previous Percutaneous Coronary Interventions (PCI) of the target lesion.
17. Previous PCI of the target vessel within 9 months pre-procedure.
18. Planned PCI of any vessel within 30 days post-procedure.
19. Surgery 30 days prior to this PCI or anticipated surgery 6-months post this PCI.
20. During the index procedure, the target lesion requires treatment with a device other than PTCA prior to use of Danubio (including but not limited to cutting balloon, any atherectomy, any laser, thrombectomy, etc.).
21. Second lesion requiring treatment in target vessel.
22. Second bifurcation lesion requiring treatment.
23. History of a stroke or transient ischemic attack (TIA) within the prior 6 months.
24. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months.
25. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
26. Concurrent medical condition with a life expectancy of less than 12 months.
27. Any previous or planned treatment of the target vessel with anti-restenotic therapies including, but not limited to brachytherapy.
28. Currently participating in an investigational drug or another device trial that has not completed the primary endpoint or that clinically interferes with the current trial endpoints, or requires coronary angiography, IVUS or other coronary artery imaging procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss (mm) in Side Branche (SB) | 6 months post-procedure (up to 26 weeks)
  Late Lumen Loss at the ostium of the SB (within 5mm from the carina) by Quantitative Coronary Angiography (QCA).

SECONDARY OUTCOMES:
In-stent Late Lumen Loss (mm) in Main Branch (MB) | 6 months post-procedure (up to 26 weeks)
  In-stent Late Lumen Loss in the MB by QCA.
Angiographic Binary Restenosis rate (%) | 6 months post-procedure (up to 26 weeks)
  Angiographic binary restenosis rate (%) in the side and main branches by QCA.
Major Adverse Cardiac Event (MACE) rate | In-hospital, 1, 6 and 12 months post-procedure.
  MACE defined as death, Myocardial Infarction (MI, Q waves and non-Q waves), emergent cardiac bypass surgery, or any target lesion revascularization (repeat Percutaneous transluminal coronary angioplasty (PTCA) or Coronary artery bypass grafting (CABG)).
Clinically-driven Target Lesion Revascularization (TLR) | 1, 6 and 12 months post-procedure
Target Vessel Failure (TVF) | 1, 6 and 12 months post-procedure
Target Vessel Revascularization (TVR) | 1, 6 and 12 months post-procedure
Angiographic success | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BERLAND, MD, Principal Investigator — Clinique Saint Hilaire - ROUEN
Locations (7):
- France (7):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Pôle Santé République, Clermont-Ferrand
  - Centre Cardiologique d'Evecquemont, Évecquemont
  - Institut hospitalier Jacques Cartier, Massy
  - CHU Nantes, Nantes
  - Clinique Saint-Hilaire, Rouen
  - Clinique Pasteur, Toulouse

REFERENCES:
- [Derived] Berland J, Lefevre T, Brenot P, Fajadet J, Motreff P, Guerin P, Dupouy P, Schandrin C; DEBSIDE trial investigators. DANUBIO - a new drug-eluting balloon for the treatment of side branches in bifurcation lesions: six-month angiographic follow-up results of the DEBSIDE trial. EuroIntervention. 2015 Dec;11(8):868-76. doi: 10.4244/EIJV11I8A177. PMID 26696455